CLINICAL TRIAL: NCT00368758
Title: The Effect of Probioticson Bloating in IBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Veterinary and Agricultural University, Denmark (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: JRA1
Record Dates: First submitted 2006-08-24; First posted 2006-08-25 (Estimated); Last update posted 2006-08-25 (Estimated); Status verified 2006-08

CONDITIONS: Irritable Bowel Syndrome
Keywords: Meteorism; Bloating; Irritable bowel syndrome (IBS); Probiotics; Bowel gas
MeSH Terms: conditions — Irritable Bowel Syndrome

INTERVENTIONS:
Drug: Probiotic bacteria (Trevis R)

SUMMARY:
The purpose of the study is to establish an in-vitro method to evaluate the effect of probiotics on gas production in feces (hydrogen and methane)

DETAILED DESCRIPTION:
The objective of this study is to establish a model for screening probiotic bacteria in the treatment of meteorism symptoms (feeling of air in the stomach) with otherwise healthy adult women. As excessive bacterial gas production in the intestine is the most likely mechanism behind meteorism, we will examine eventual changes of the production of gases (hydrogen and methane) before and after administration of Trevis®. For screening of Trevis® we will apply a combination of clinical examination and a laboratory model for the determination of gastrointestinal gas production (a new method in connection with studies on probiotics). The results will be compared with the test person's specification of their health, both with respect to gastrointestinal function and in general through questionnaires. The background for the project will be described in the following.

ELIGIBILITY:
Inclusion Criteria:

- Female test persons with symptoms of meteorism, the age of > 18 years, completely integrated in the Danish society (including nutrition), and no previous abdominal surgery besides from appendicectomy (advertisement in a local newspaper for test persons).

Exclusion Criteria:

* Lactose and sorbitol intolerant persons (based on hydrogen breath tests).
* Persons with chronic ingestion of medicine, that might have an effect on gut bacterial flora or bowel motility.
* Persons taking antibiotics within 2 month prior to the trial
* Persons with diagnosed gastrointestinal disease other than IBS.
* Persons not able to understand and/or read Danish.
* Persons under age and persons with obvious problems remembering and sticking to the protocol (persons with dementia, psychological illness etc.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-08; Study Completion 2007-09

PRIMARY OUTCOMES:
In-vitro production (quantified) of hydrogen and methane in feces
Recovery of ingested bacteria in feces by PCR

SECONDARY OUTCOMES:
Quality of life (SF36-danish version)
VAS-scores for bloating, distention, abdominal pain, abdominal discomfort, flatulence
Abdominal height in lying position, waist circumference, weight

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Andersen, MD, Principal Investigator — Dept. Human Nutrition, The Royal Veterinary and Agricultural University, Copenhagen
Locations (1):
- Dept. Human Nutrition, The Royal Veterinary and Agricultural University, Copenhagen, Denmark

REFERENCES:
- [Background] Strocchi A, Levitt MD. Factors affecting hydrogen production and consumption by human fecal flora. The critical roles of hydrogen tension and methanogenesis. J Clin Invest. 1992 Apr;89(4):1304-11. doi: 10.1172/JCI115716. PMID 1556190